CLINICAL TRIAL: NCT05743023
Title: Evaluation of an Ayurvedic Whole Systems-based Lifestyle Protocol for Quality of Breast Cancer Survivorship: A Randomized Controlled Pilot Study
Brief Title: Consciousness-based Ayurveda Lifestyle Program for Improving Quality of Life in Survivors of Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Robert Schneider, MD (Other)
Responsible Party: Sponsor-Investigator, Robert Schneider, MD, Director, Institute for Natural Medicine and Prevention; Dean, College of Integrative Medicine, Maharishi International University
Organization: Maharishi International University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 07102022_SR
Record Dates: First submitted 2022-10-25; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer Survivors
Keywords: Breast cancer; Breast cancer survivorship; Ayurveda; Lifestyle; Integrative; Mind-body medicine
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consciousness-based Ayurvedic lifestyle Intervention (Experimental): In the intervention group, each participant will receive a structured education and be asked to follow a 12-week personalized diet and daily routine protocol based on the assessment of their current Ayurvedic mind-body state. Participants will be asked to complete the self-reported questionnaires at baseline, 6, and 12-week.
  Interventions: Behavioral: Ayurvedic lifestyle protocol
- Waitlist control (Active Comparator): Participants in the waitlist control group will not receive any intervention. They will continue usual care and will be asked to complete the self-reported questionnaires at baseline, 6, and 12-week. Participants n this group receive their personalized protocol at the end of 12 weeks after completing all the data collection.
  Interventions: Behavioral: Ayurvedic lifestyle protocol

INTERVENTIONS:
Behavioral: Ayurvedic lifestyle protocol — Based on each participant's current mind-body imbalance determination, a personalized 12-week intervention lifestyle protocol will be given.
  Each protocol will mainly address diet and daily routine, quality of food, food combinations, and living in harmony with natural rhythm for balancing the predominant imbalance based on Ayurvedic principles. In addition, the lifestyle protocol will also include stress-reducing methods and more specifically, participants will be recommended to learn and practice the Transcendental Meditation technique.
  Other Names: personalized diet and daily routine protocol

SUMMARY:
This study is a pilot study to assess the feasibility and effectiveness of a 12-week intervention of personalized diet and lifestyle protocol based on the principles of Ayurveda's whole systems approach to achieving improvement in a) quality of life, b) digestive health, c) sleep among women breast cancer survivors.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among women worldwide. Due to advancements in early diagnosis and treatment, the survival rate of breast cancer has significantly increased. According to the National Cancer Institute's office of cancer survivorship, as of January 2019, there are 3.8 million breast cancer survivors.

Evidence indicates that cancer survivors experience many adverse effects of treatment and suffer from significant quality of life (QOL) challenges such as depression, anxiety, emotional, social, psychological, physiological, and spiritual wellbeing.

Personalized diet, lifestyle and daily routine approaches to breast cancer survivorship are often undervalued. Generally, the dietary guidelines are based only on an individual's nutritional and caloric needs.

Due to the increasing number of breast cancer survivors, it has become essential to have evidence-based guidelines for breast cancer survivorship to improve digestive health, QOL, and general wellbeing. Understanding the science behind personalized lifestyle-related factors, including diet, exercise, and emotional and spiritual wellbeing in cancer survivorship, is urgently needed. Digestive health and the gut microbiome may play an important role in the QOL after surviving breast cancer; however, there are fewer studies on the relationship between diet and daily routine to gut health and breast cancer survivorship care.

This study will test whether personalized guidelines based on the principles of Maharishi Ayurveda - a whole systems approach to reducing strength, improving digestive health and living in harmony with the circadian rhythm to improve QOL for women diagnosed and treated for breast cancer. In addition to that, this pilot study may provide preliminary data to further develop a clinical practice guideline that is cost-effective and easy to follow for women breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* A breast cancer survivor in remission (Females ≥ 18 years)
* Diagnosis of stage I-IV breast cancer
* Three months or more after receiving conventional treatment (chemotherapy, radiation therapy, and/or surgery)
* Willing to comply with the study intervention recommendations for 12 weeks
* English speaking
* Have access to technology to participate in zoom visits

Exclusion Criteria:

* Male responders
* Inability to provide informed consent
* Physiological or psychological debility that would interfere with the ability to participate in the study fully
* Active metastatic or recurrent disease (to avoid early withdrawal from the study)
* Anticipates undergoing surgery during the duration of the intervention
* Substance abuse (to avoid early withdrawal from the study)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of life | 0, 6 weeks, and 12 weeks
  Assess change from baseline quality of life to 6 and 12 weeks.
  Researchers will use the following Self-reported outcome measure instruments:
  Quality of life: Quality of Life instrument (cancer patient/cancer survivor version) developed by the City of Hope National Medical Center in California.
Change in Digestive health | 0, 6 weeks, and 12 weeks
  Assess change from baseline digestive health to 6 and 12 weeks.
  Researchers will use the following Self-reported outcome measure instruments:
  Ayurvedic assessment of digestive strength questionnaire and Gastrointestinal Symptoms Rating Scale (GSRS) for the gut health assessment.
Change in Sleep disturbance | 0, 6 weeks and 12 weeks
  Assess change from baseline sleep disturbance to 6 and 12 weeks.
  Researchers will use the following Self-reported outcome measure instruments:
  Assessment using the General Sleep Disturbance Scale (GSDS).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schneider, MD, Principal Investigator — Maharishi International University, Fairfield, Iowa
Locations (1):
- Maharishi International University, Richmond, California, United States